CLINICAL TRIAL: NCT06274931
Title: Analysis of the Pulmonary Microbiome
Status: Recruiting | Type: Observational
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Andrea Bruni, Professor, University Magna Graecia
Other Study IDs: 373
Record Dates: First submitted 2024-02-01; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Pneumonia; Microbial Colonization; Microbial Disease
MeSH Terms: conditions — Pneumonia; Communicable Diseases | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bronchoalveolar lavage (BAL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ICU patients: Patients admitted to the Intensive Care Unit with a diagnosis of acute respiratory failure
  Interventions: Procedure: Bronchoscopy
- non ICU patients: Outpatient patients with a diagnosis of pneumonia
  Interventions: Procedure: Bronchoscopy
- Controls: In the control group, an alveolar bronchial lavage was performed directly on lung tissue taken from deceased individuals who did not have any known lung pathologies.

INTERVENTIONS:
Procedure: Bronchoscopy — Through a bronchoscopic examination performed at the time of admission for diagnostic purposes, an alveolar bronchial lavage was performed for the analysis of the lung microbiome.
  Groups: ICU patients; non ICU patients

SUMMARY:
The purpose of the protocol is to study the pulmonary microbiome in patients who develop pneumonia.

DETAILED DESCRIPTION:
The purpose of the protocol is to study the pulmonary microbiome in patients who develop pneumonia with severe acute respiratory failure, requiring admission to the Intensive Care Unit, and to compare it with that of patients diagnosed with pneumonia but who do not develop severe acute respiratory failure and subsequent admission to the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute respiratory failure
* Patients with suspect of pneumonia

Exclusion Criteria:

* pregnancy
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of three groups: one ICU-patients with a diagnosis acute respiratory failure, another group of non - ICU patients, and finally, a control group of individuals without pulmonary involvement.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of Lung Microbiome in Acute Respiratory Failure | The study will be conducted over a period of two months, during which data collection, bronchoscopic examinations, and analysis of the lung microbiome will be carried out.
  This study aims to investigate the composition and diversity of the lung microbiome in patients experiencing acute respiratory failure. Specifically, the research evaluates differences in the lung microbiome between ICU-admitted patients, non-hospitalized individuals, and a control group without known lung pathologies. Through bronchoscopic examinations and alveolar bronchial lavage, the study seeks to elucidate potential associations between lung microbiota and the development of acute respiratory failure. For the analysis of the lung microbiome, the MiSeq Reagent Nano v2 kit is utilized. This kit enables high-throughput sequencing of microbial DNA extracted from samples obtained via bronchoscopic examinations and alveolar bronchial lavage. The MiSeq platform provides accurate and comprehensive data on the microbial composition and diversity present in the lung microbiome of study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bruni, Principal Investigator — Magna Graecia University
Locations (1):
- University Hosp[ital, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No